CLINICAL TRIAL: NCT02602613
Title: AMEND I Study - for the Valcare Medical AMEND TM Mitral Valve Repair System
Brief Title: AMENDTM Mitral Valve Repair System, Annuloplasty Ring Applied in a Transcatheter Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valcare Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL4-0001P
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2017-10

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

ARMS (1):
- AMEND (Experimental)
  Interventions: Device: AMEND Mitral Valve Repair System

INTERVENTIONS:
Device: AMEND Mitral Valve Repair System — Annuloplasty ring applied in a transcatheter method

SUMMARY:
A multi center study to evaluate the safety of the AMENDTM Mitral Valve Repair System and its ability to reduce mitral regurgitation. AMEND device is an annuloplasty ring implanted in a minimally invasive trans-catheter method.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥18
* The patient requires mitral valve annuloplasty for mitral regurgitation without the need for concomitant cardiovascular surgical procedures
* NYHA functional capacity ≥2
* The subject is high risk to undergo a mitral valve surgery as assessed by the center heart team
* The patient is willing to comply with study procedures and is available to return to the implant center for follow-up visits.
* The patient is willing to provide Informed consent

Exclusion Criteria:

* Cardiac or non-cardiac major or progressive disease, which in the investigator's discretion produces an unacceptable increased risk to the patient.
* Life expectancy of less than twelve months.
* Heavily calcified annulus or leaflets.
* Previous or active endocarditis.
* Active infection.
* A previously implanted prosthetic mitral valve or annuloplasty ring/band.
* The patient is contraindicated to general anesthesia.
* Pregnant (urine HCG test result positive) or lactating patient.
* Drug or alcohol abuse.
* Participation in concomitant research studies of investigational products that will interfere with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Safety - Freedom from major SAE's at 30 days following procedure | 30 days
  Freedom from major SAE's at 30 days following procedure
Technical success of implantation | End of procedure
  Ring location and attachment based on echocardiography

SECONDARY OUTCOMES:
Safety - Freedom from major SAE's at 6 months following procedure | 6 months
  Freedom from major SAE's at 6 months following procedure

CONTACTS AND LOCATIONS:
Locations (5):
- ZNA Middelheim Hospital, Antwerp, Belgium
- Na Homolce Hospital, Prague, Czechia
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Azienda Ospedaliera Di Padova, Padua, Italy